CLINICAL TRIAL: NCT00559182
Title: A Phase I Dose Escalation Study of MK-8033 in Patients With Advanced Solid Tumors
Brief Title: A Study of MK-8033 in Patients With Advanced Solid Tumors (MK-8033-001)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 8033-001; 2007_590
Record Dates: First submitted 2007-11-14; First posted 2007-11-16 (Estimated); Last update posted 2022-07-26 (Actual); Status verified 2022-07

CONDITIONS: Advanced Cancer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Parts A and B: MK-8033 (Experimental): Dose Escalation Study
  Interventions: Drug: Comparator: MK-8033
- Part C: MK-8033 +/- omeprazole (Experimental): Crossover Study
  Interventions: Drug: Comparator: MK-8033 +/- omeprazole

INTERVENTIONS:
Drug: Comparator: MK-8033 — MK-8033 will be administered as an oral formulation in sequentially rising dose levels starting at 50 mg and continuing at 100% dose increments until dose level 4 (800 mg total daily dose). Dose levels 5 to 11 will be escalated at ~40% dose increments until 3000mg (total daily dose). The daily dose of MK-8033 will be divided into two equal doses. MK-8033 will be administered in a first cycle of 14 days (continuous drug administration from Day 1 through Day 14), followed by a 1 week drug holiday (Cycle 1, Day 15 through Day 21). Subsequent cycles of MK-8033 will be administered for 14 days (Cycles 2 to 4) and 28 days (Cycle 5 and beyond).
  Enrollment in Parts A and B has been completed.
  Arms: Parts A and B: MK-8033
Drug: Comparator: MK-8033 +/- omeprazole — Part C will occur at only one of the investigational sites.
  In Cycle 1, patients will be randomized to one of two treatment sequences, A/B or B/A, over two treatment periods. Treatment A: 770 mg MK-8033 twice daily with co-administration of 20 mg omeprazole once daily. Treatment B: 770 mg MK-8033 twice daily. After Cycle 1 is complete, patients may continue to receive MK-8033 until disease progression or unacceptable toxicity.
  Enrollment for Part C has been suspended.
  Arms: Part C: MK-8033 +/- omeprazole

SUMMARY:
This is a first-in-human trial to establish the safety, tolerability, Recommended Phase II Dose (RP2D), pharmacodynamic, and clinical activity of MK-8033.

Parts A and B of the study will determine the maximum tolerated dose (MTD) and RP2D. Part C of the study will be a single panel crossover study to determine the effect of omeprazole, a gastric pH modifier, on the pharmacokinetics of MK-8033.

ELIGIBILITY:
Inclusion Criteria:

* Patient must be at least 18 years of age, with adequate organ function, and an Eastern Cooperative Oncology Group (ECOG) performance of <2
* Patient must be willing to undergo pre-study and post-dose tumor biopsy and have tumor accessible for biopsy (Waived during Parts A and C)

Exclusion Criteria:

* Patient is currently using bisphosphonate therapy or has received this therapy in past 6 months
* Patient has had chemotherapy, radiotherapy, or biological therapy within 4 weeks of study participation
* Patient has history of cardiac disease
* Patient with a primary central nervous system tumor
* Patient has a known psychiatric or substance abuse disorder
* Patient is pregnant or breastfeeding, or expecting to conceive during the study
* Patient is known to be Human Immunodeficiency Virus (HIV) positive and the HIV infection is not well controlled
* Patient has received therapy with a Proton-Pump Inhibitor, Histamine2-Receptor antagonist or antacid within one week of study participation (Part B only)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2007-12-05 (Actual); Primary Completion 2010-06-10 (Actual); Study Completion 2010-07-09 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of MK-8033 based on drug-related dose limiting toxicity. | for the entire duration of study (27 months)
Recommended Phase II Dose (RP2D) based on safety, tumor pharmacodynamics, and pharmacokinetics | for the entire duration of study (27 months)
Plasma area under the curve (AUC) for F2 formulation alone or in combination with omeprazole | Day 1-21
Safety and tolerability of MK-8033 F2 formulation alone or in combination with omeprazole based on incidence of adverse experiences | Day 1-21
Tumor Pharmacodynamics (PD): phospho-c-Met (MET or MNNG HOS Transforming gene) Levels (Parts A & B) | Cycle 1 pre-dose & Day 12
Tumor PD: phospho-Akt (Protein Kinase B) Levels (Parts A & B) | Cycle 1 pre-dose & Day 12
Tumor PD: phospho-MAPK (mitogen-activated protein kinase) Levels (Parts A & B) | Cycle 1 pre-dose & Day 12
Bone PD: Cross-Linked N-telopeptides of Type I collagen (NTx) Levels (Parts A & B) | Baseline, Cycle 1 Day 8, & Cycle 3 Day 1

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- [Result] Keedy VL, Lenz HJ, Saltz L, Whisenant JG, Berlin JD, Camacho LH. First-in-human phase I dose escalation study of MK-8033 in patients with advanced solid tumors. Invest New Drugs. 2018 Oct;36(5):860-868. doi: 10.1007/s10637-018-0567-z. Epub 2018 Jan 29. PMID 29376210